CLINICAL TRIAL: NCT04953975
Title: Association of Functional Dyspepsia Symptom Diary Score and Other Scores Related to Functional Dyspepsia and Its Severity
Status: Completed | Type: Observational
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Associated professor, Air Force Military Medical University, China
Other Study IDs: KY20202087-F-2
Record Dates: First submitted 2021-06-29; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: Functional Dyspepsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Functional dyspepsia (FD) is a common functional gastrointestinal disease. Several patient-reported outcome questionnaires have been established to evaluate the severity of FD, including Dyspepsia Symptom Severity Index (DSSI), Nepean Dyspepsia Index (NDI), and Short-Form Nepean Dyspepsia Index (SF-NDI). Functional Dyspepsia Symptom Diary (FDSD) is a newly symptom-focused patients-reported outcome measure raised by the Patient-Reported Outcome Consortium's Functional Dyspepsia Working Group. The association of the novel FDSD and other scores-related to FD has not been fully investigated. Furthermore, the severity of FD is varied among different patients. It remains unclear how the moderate and severe FD can be defined by the FDSD.

ELIGIBILITY:
Inclusion Criteria:

* 1. 18-70 years old
* 2. Patients who met the Rome IV diagnostic criteria of FD
* 3. Normal upper endoscopy and abdominal ultrasonography within one year.

Exclusion Criteria:

* 1, Patients with local or systemic diseases which may cause dyspeptic symptoms:

  1. Known active peptic ulcer, cholecystitis, gallstone, gastrointestinal obstruction, gastroparesis, and etc.
  2. Known acute or chronic diseases of liver or kidney
  3. Obvious hematological abnormality, or endocrine and metabolic diseases
  4. suspected incomplete or complete bowel obstruction
  5. Known malignancy
  6. Other conditions which may be associated with dyspeptic symptoms (such as NSAIDs associated dyspepsia)
* 2, Pregnancy
* 3, Inability to give informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18-70 years old who met the Rome IV diagnostic criteria of FD with normal upper endoscopy and abdominal ultrasonography within one year were eligible for our study. Patients with local or systemic diseases which may cause dyspeptic symptoms were excluded. Patients who were pregnant or unable to give informed consent were also excluded.
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-06-20 (Actual); Study Completion 2021-06-20 (Actual)

PRIMARY OUTCOMES:
Functional Dyspepsia Symptom Diary | 1 day
  The FDSD consists of 5 cardinal items (burning in the stomach, stomach pain, bloating, postprandial fullness, and early satiety) and 3 supplementary items (nausea, burping/belching rating, and burping/belching bother). Each item can be scored from 0 (no) to 10 (worst). Total Symptom Score includes the 5 cardinal items and ranges from 0 to 50.

SECONDARY OUTCOMES:
Gastrointestinal Symptom Rating Scale (GSRS) | 1 day
  The GSRS contains 15 items. All individual items are scored on a 7-point Likert scale (1 = not at all to 7 = extremely) and are subsequently clustered into five domains (abdominal pain, reflux, indigestion, diarrhea, and constipation); higher scores indicate more severe symptoms.
Dyspepsia Symptom Severity Index (DSSI) | 1 day
  The DSSI contains 20 items. All individual items are scored on a 5-point Likert scale (0 = not at all to 4 = extremely) and are subsequently clustered into three domains (Dysmotility-like, Reflux-like, and Ulcer-like); higher scores indicate more severe symptoms.
Short Form of Nepean Dyspepsia Index (SF-NDI) | 1 day
  The SF-NDI consists of 10 questions regarding the effects of dyspepsia symptoms ("stomach problems") on different aspects of life (tension, interference with daily activities, eating/drinking, knowledge/control, and work/study). Each response can be from 1 (not at all affected) to 5 (extremely affected), or 0 (N/A), for a total summed score out of 50.
Hamilton Anxiety and Depression Scale | 1 day
  Anxiety and depression of patients are assessed by using Hamilton Anxiety and Depression Scale.
Severity of FD judged by patients | 1 day
  Patients were asked to rate the severity of FD as mild, moderate, and severe.
Severity of FD judged by physicians | 1 day
  Physicians rated the patients' severity of FD as mild, moderate, and severe.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi

REFERENCES:
- [Derived] Shi X, Luo H, Wang X, Ren G, Zhang L, Tao Q, Liang S, Liu N, Huang X, Zhang X, Deng H, Qin W, Kang X, Pan Y, Fan D. Functional dyspepsia symptom diary is correlated with other questionnaires and associated with severity in patients with functional dyspepsia: a multicenter, prospective observational study. J Gastroenterol Hepatol. 2022 Jul;37(7):1298-1306. doi: 10.1111/jgh.15854. Epub 2022 Apr 23. PMID 35434810